CLINICAL TRIAL: NCT03340506
Title: Open Label, Multi-center Roll-over Study to Assess Long Term Safety in Patients Who Have Completed a Global Novartis or GSK Sponsored Dabrafenib and/or Trametinib Study
Brief Title: Dabrafenib and/or Trametinib Rollover Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDRB436X2X02B; 2023-509318-13-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Melanoma; Non Small Cell Lung Cancer; Solid Tumor; Rare Cancers; High Grade Glioma
Keywords: Tafinlar; Mekinist; Dabrafenib; Trametinib; Adult; Melanoma; Melanoma Stage IV; Metastatic Melanoma; Advanced Melanoma; Lung Cancer; NSLC; Non Small Cell Lung Cancer; BRAF V600 Mutation; BRAF Gene Mutation; Solid tumor; Rare cancers; High Grade Glioma
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Glioma; Lung Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- dabrafenib monotherapy (Experimental): Patients in this study may receive:
  - monotherapy of dabrafenib
  Interventions: Drug: dabrafenib
- trametinib monotherapy (Experimental): Patients in this study may receive:
  - monotherapy of trametinib
  Interventions: Drug: trametinib
- Combination therapy (dabrafenib & trametinib) (Experimental): Patients in this study may receive:
  - the combination of dabrafenib and trametinib
  Interventions: Drug: dabrafenib; Drug: trametinib

INTERVENTIONS:
Drug: dabrafenib — dabrafenib is available in capsules (50mg and 75mg) taken twice a day
  Arms: Combination therapy (dabrafenib & trametinib); dabrafenib monotherapy
Drug: trametinib — trametinib is available in tablets (0.5mg, 2mg dose)
  Arms: Combination therapy (dabrafenib & trametinib); trametinib monotherapy

SUMMARY:
This study is to provide access for patients who are receiving treatment with dabrafenib and/or trametinib in a Novartis-sponsored Oncology Global Development, Global Medical Affairs or a former GSK-sponsored study who have fulfilled the requirements for the primary objective, and who are judged by the investigator as benefiting from continued treatment in the parent study as judged by the Investigator at the completion of the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently receiving treatment with dabrafenib/trametinib monotherapy or combination within a Novartis or former GSK sponsored study which has fulfilled the requirements for the primary objective.
* In the opinion of the Investigator would benefit from continued treatment.

Exclusion Criteria:

* Patient has been previously permanently discontinued from study treatment in the parent protocol.
* Patient's indication is commercially available and reimbursed in the local country.
* Patient currently has unresolved toxicities for which dabrafenib and/or trametinib dosing has been interrupted in the parent study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-28 (Actual); Primary Completion 2029-12-18 (Estimated); Study Completion 2030-12-28 (Estimated)

PRIMARY OUTCOMES:
Occurences of adverse events to evaluate long term safety and tolerability of dabrafenib, trametinib or combination | Baseline up to approximately 10 years after the first subject's first visit, or will remain open until treatment becomes commercially available and reimbursed, or another access program becomes available, whichever comes first.
  Clinical and laboratory assessments should be completed based on the local standard of care and physician practice for routine safety monitoring. More frequent examinations may be performed at the Investigator's discretion if medically indicated. Any abnormalities considered clinically significant, induce clinical signs or symptoms, or require changes in treatment constitute an adverse event.

SECONDARY OUTCOMES:
Clinical Benefit Assessment by investigator | Baseline up to approximately 10 years after the first subject's first visit, or will remain open until treatment becomes commercially available and reimbursed, or another access program becomes available, whichever comes first.
  To evaluate clinical benefit as assessed by the Investigator

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- United States (4):
  - Honor Health Research Institute, Scottsdale, Arizona
  - National Institute Of Health, Bethesda, Maryland
  - James Cancer Hospital and Solove Research Institute Ohio State, Columbus, Ohio
  - Mary Crowley Cancer Research, Dallas, Texas
- Novartis Investigative Site, Caba, Buenos Aires, Argentina
- Novartis Investigative Site, Innsbruck, Tyrol, Austria
- Novartis Investigative Site, Beijing, China
- Novartis Investigative Site, Copenhagen, Denmark
- France (4):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Germany (4):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
- Hungary (2):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
- Japan (2):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Chuo Ku, Tokyo
- Netherlands (2):
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Utrecht
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Songkhla, Hat Yai, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com